CLINICAL TRIAL: NCT00825175
Title: The Effect of Treadmill Training and Orthotic Use on the Development of Walking and Upright Play in Infants With Down Syndrome
Brief Title: Treadmill Training and Orthotic Use in Infants With Down Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Julia Looper, Graduate Student, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00002466
Record Dates: First submitted 2009-01-15; First posted 2009-01-19 (Estimated); Results first posted 2014-01-24 (Estimated); Last update posted 2017-12-04 (Actual); Status verified 2017-10

CONDITIONS: Down Syndrome
Keywords: Down syndrome; Gait; Motor Development; Orthoses
MeSH Terms: conditions — Down Syndrome | interventions — Orthotic Devices; Braces

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Treadmill Training in infants with Down syndrome only
  Interventions: Behavioral: Treadmill Training
- 2 (Experimental): Treadmill Training and supramalleolar orthoses use for infants with Down syndrome
  Interventions: Behavioral: Treadmill Training; Device: Supramalleolar Orthoses

INTERVENTIONS:
Behavioral: Treadmill Training — Parents hold their infants on an infant treadmill for 8 minutes a day, 5 days a week. The treadmill speed is set at 0.2 m/s.
Device: Supramalleolar Orthoses — In addition to treadmill training the infants receive Supramalleolar orthoses. They wear the orthoses for 8 hours a day, 5 days a week.
  Other Names: Orthoses; Orthotics
  Arms: 2

SUMMARY:
This study determines the effect of orthotic use in combination with treadmill training on the development of gross motor skills and walking onset in infants with Down syndrome.

DETAILED DESCRIPTION:
The goal of this study is to determine if orthotic use impacts the development of walking and upright play skills over and above the impact that treadmill training alone has. Infants with Down syndrome who can pull to stand but not walk will be recruited and assigned to a group that receives treadmill training and orthoses or just treadmill training. The infants are followed monthly until they have one month of walking experience. During the monthly visits, the infants' gross motor development is tested and their upright play behavior is observed. At the end of the study each infants gait is evaluated. We believe that the orthoses will lead to a decreased age at walking onset, an improvement in gait patterns, and an improvement in upright play ability.

ELIGIBILITY:
Inclusion Criteria:

* Trisomy 21
* Able to pull to stand but not walk

Exclusion Criteria:

* Additional developmental diagnoses
* Uncorrected vision or hearing impairments
* Previous orthotic intervention
* Previous treadmill intervention

Ages: 6 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2006-03; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julia Looper, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] Looper J, Ulrich DA. Effect of treadmill training and supramalleolar orthosis use on motor skill development in infants with Down syndrome: a randomized clinical trial. Phys Ther. 2010 Mar;90(3):382-90. doi: 10.2522/ptj.20090021. Epub 2010 Jan 14. PMID 20075148

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment in Winter 2007 for in home intervention.
Pre-assignment Details: Subjects were excluded if they previously had worn foot orthoses
Groups:
- Treadmill Training Only: This group received treadmill training in home for 8 min per day/ 5 days per week. Training started when the children pulled to stand and ended when they could take 3 independent steps.
- Treadmill Training and Orthotic Use: This group received treadmill training from the time they could pull to stand until they could take 3 independent steps. They also work supramalleolar foot orthoses for 8 hours a day during that time frame.
Period: Overall Study
Arm/Group | Treadmill Training Only | Treadmill Training and Orthotic Use
Started | 10 | 12
Completed | 10 | 7
Not Completed | 0 | 5
Not completed — Withdrawal by Subject | 0 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treadmill Training Only | Treadmill Training and Orthotic Use | Total
Number analyzed (Participants) | 10 | 12 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10 | 12 | 22
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 12 (2) | 12 (2) | 12 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 6 | 7 | 13
Region of Enrollment [Number; unit: participants]
  United States | 10 | 12 | 22

OUTCOME MEASURES:

1. Primary Outcome: Pattern of Gross Motor Development
Description: Age in months at walking development as indicated by the Gross Motor Function Measure, a standardized test of gross motor development.
Time Frame: monthly; starting when child can pull to stand and ending when the test determined that the child was walking.
Population: analysis was on protocol
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Treadmill Training Only | Treadmill Training and Orthotic Use
Number analyzed (Participants) | 10 | 7
months | 28.2 (8.3) | 28.3 (5.9)

ADVERSE EVENTS:
Arm/Group | Treadmill Training Only | Treadmill Training and Orthotic Use
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/12
Other Adverse Events (participants affected / at risk) | 0/10 | 0/12

LIMITATIONS AND CAVEATS:
small sample size

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes